CLINICAL TRIAL: NCT02743481
Title: Early Life Exposures in Agriculture
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916095; 16-C-N095
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Testicular Cancer; Leukemia; Lymphoma; Brain Cancer
Keywords: Pesticide; Agriculture; Cancer; Childhood; Leukemia
MeSH Terms: conditions — Testicular Neoplasms; Leukemia; Lymphoma; Brain Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

The Agricultural Health Study (AHS) studied farmers and their spouses in North Carolina and Iowa. It also included people who worked with pesticides in Iowa. They answered a questionnaire and gave data about their children born since 1975. Researchers want to link this data to public data like birth and death certificates. They want to study how early life exposures to farms are linked to cancer and other bad health outcomes.

Objective:

To study data to find links between early life farm exposure and negative health outcomes.

Eligibility:

There will be no human subjects.

Design:

Researchers will get public data in the two study states. This will come from things like:

Birth certificates

Driver s licenses

Voter registration

Death certificates

Based on these plus the AHS data, they will create a study group. It will be called Early Life Exposure in Agriculture (ELEA).

Researchers will link ELEA data to cancer data. This will identify prevalence of cancer.

They will study parents answers on the AHS. The topics include farm practices and pesticide use. They will determine ELEA exposure to pesticides.

Researchers will analyze the cancer and pesticide results and look for links.

DETAILED DESCRIPTION:
There is increasing evidence that early life exposures may influence future health outcomes although there is a critical need to more fully understand how these may differ from exposures received later in life. The farm environment includes pesticides that have been suggested to increase cancer risk in both children and adults. A review of the literature identified crucial gaps in our knowledge and highlighted the need for accurate exposure assessment, including separate parental interviews, specific pesticide exposure questions, and semiquantitative exposure measures that can be used to confirm information obtained through questionnaires 2. Some studies suggest that the timing of exposure may be particularly important. For example, in a study of the insecticide DDT and breast cancer, researchers observed the highest risks among women exposed prior to age 14 compared to later in life 3. The agricultural environment also includes other exposures such as animals, allergens, and endotoxins. These exposures may influence immune function, particularly when exposed at a young age, and subsequently affect later cancer risk.

The Agricultural Health Study (AHS) is a prospective cohort study of farmers and their spouses residing in North Carolina and Iowa, and commercial pesticide applicators residing in Iowa. At enrollment (1993-7) women (farmers and spouses of farmers) provided information on their children born since 1975, including name, gender, SSN and dates of birth. In previous analyses conducted using Iowa AHS data only for cancer incidence and all-cause mortality in children under the age of 19, findings suggested increased risks of incident cancer among these children associated with the use of certain pesticides by their parents. The mortality analysis focused on fatal injuries sustained, indicative of the dangerous nature of working on the farm6. In collaboration with researchers at the University of Iowa, we are currently updating the previous analysis with new cancer incidence information through 2011 and information provided by the University of Iowa, which has performed a linkage to Iowa birth certificates to identify additional children born to AHS participants from 1975-2009.

With this proposal, we are proposing to further expand the linkages in Iowa to include children not previously included, and to link to the North Carolina registries for the first time to identify additional 2 births, cancer incidence and mortality. This will establish a unique cohort of agriculturally exposed offspring, with comprehensive information on their parents farming practices, as well as other information. These data will be used to evaluate the hypothesis that early life agricultural exposures influence cancer risk. Previous analyses have only focused on childhood cancers; we will include cancers diagnosed from birth through adulthood.

ELIGIBILITY:
* INCLUSION CRITERIA:
* children born to Agricultural Health Study (AHS) participants from 1975-2009.
* individuals identified through questionnaire or through the probabilistic and deterministic match to the birth registries as being the offspring of the AHS participants.

Ages: 7 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Offspring of Agricultural Health Study (AHS) cohort members (farmers and their spouses residing in North Carolina and Iowa, and commercial pesticide applicators residing in Iowa).
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Cancer incidence | Birth through 2014
  Cancer incidence
Mortality | Birth through 2014
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beane-Freeman, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States